CLINICAL TRIAL: NCT01123239
Title: Reducing Racial Disparities in Diabetes Care - The Coached Care Study
Brief Title: Understanding and Improving Diabetes Care for Ethnic Minorities
Acronym: R2D2C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sheldon Greenfield, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS# 2004-4025; R18DK069846 (NIH); K01DK078939 (NIH)
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Healthcare Disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coached Care (Experimental): Coached Care pairs patients with linguistically and ethnically matched peer "coaches" who have been trained to promote patient participation in the medical visit. The coaches, who themselves have diabetes, meet with patients immediately before each of their regularly scheduled medical visits to encourage active involvement in information seeking and decision-making.
  Interventions: Behavioral: Coached Care
- Standard Diabetes Education (Active Comparator): Patients receive one-on-one diabetes education sessions before each medical visit. These sessions are purely informational, and do not include the specific patient activation components of the coached care intervention.
  Interventions: Behavioral: Standard Diabetes Education

INTERVENTIONS:
Behavioral: Coached Care — Coached Care pairs patients with linguistically and ethnically matched peer "coaches", who themselves have diabetes, and have been trained to meet with patients immediately before each of their regularly scheduled medical visits to encourage active involvement in information seeking and decision-making. Using a decision tree algorithm, they help patients identify relevant questions about symptoms, barriers to self-management and treatment options to discuss with doctor. They encourage mutual decision-making about tailoring the patient's medication regimen, diet and physical activities and work with the patients to overcome barriers to communication with their doctor. After the medical visit, the coach and patient review any treatment decisions and goals for self-care.
  Arms: Coached Care
Behavioral: Standard Diabetes Education — Patients randomized to the control group will receive 20 minutes of standardized diabetes education delivered by staff research assistants. Education materials have been adapted from materials developed by the American Diabetes Association. The content of these materials includes information about the causes and complications of diabetes, as well as ways to reduce complication risks. Patients in the control arm will receive 20 minutes of standardized diabetes education before each visit
  Arms: Standard Diabetes Education

SUMMARY:
In this study, we are testing the effectiveness of an intervention known as "Coached Care" to improve health outcomes and quality of care of patients being treated for type 2 diabetes, particularly patients in underserved populations. The intervention involves training members of minority communities who have diabetes to be "coaches", teaching minority patients the skills needed to participate effectively in care during office visits, as they present for those visits. Coaches follow patients for 9 routine consecutive visits, reinforcing participation skills before and between their routine office visits.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes
* At least one Hemoglobin A1c value greater than 7.5% in the year prior to recruitment.

Exclusion Criteria:

* Age above 80 years
* patients with dementia or other serious mental health problems that would prevent them from participating in the intervention.
* patients with other serious medical problems that would prevent them from participating in the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2006-01; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 1 year and 2 year follow-up
  A laboratory measure of blood sugar control

SECONDARY OUTCOMES:
Health-related quality of life | 1 year and 2 year follow-up
  Patient reported general and diabetes-specific measures of quality of life, including SF-36, diabetes burden and others.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mary and Dick Allen Diabetes Center at Hoag Hospital, Newport Beach, California
  - University of California Irvine Medical Center, Orange, California
  - Westminster Medical Center, Westminster, California

REFERENCES:
- [Derived] Malik S, Billimek J, Greenfield S, Sorkin DH, Ngo-Metzger Q, Kaplan SH. Patient complexity and risk factor control among multimorbid patients with type 2 diabetes: results from the R2D2C2 study. Med Care. 2013 Feb;51(2):180-5. doi: 10.1097/MLR.0b013e318273119b. PMID 23047130
- [Derived] Sorkin DH, Ngo-Metzger Q, Billimek J, August KJ, Greenfield S, Kaplan SH. Underdiagnosed and undertreated depression among racially/ethnically diverse patients with type 2 diabetes. Diabetes Care. 2011 Mar;34(3):598-600. doi: 10.2337/dc10-1825. Epub 2011 Jan 27. PMID 21273497
- See also: Homepage for the Reducing Racial Disparities in Diabetes Coached Care Study at UCI — http://www.medicine.uci.edu/r2d2c2/